CLINICAL TRIAL: NCT01136057
Title: A Pilot Study for Collection of High-Titer Anti-Influenza A Plasma
Brief Title: Blood and Plasma Collection For Use in Future Clinical Trials
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IDCRP-046
Record Dates: First submitted 2010-05-14; First posted 2010-06-03 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Influenza A Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be collected from participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Influenza A Exposure: Participants will include people who have recovered from influenza, received a seasonal influenza vaccine, or have both recovered from influenza and received a seasonal influenza vaccine.
  Interventions: Biological: Collection of Anti-Influenza A Immune Plasma

INTERVENTIONS:
Biological: Collection of Anti-Influenza A Immune Plasma

SUMMARY:
Treatment options are limited for the treatment of influenza. This study will collect blood from people who have been exposed to the influenza virus or who have received a seasonal influenza vaccine. The blood plasma will be used in a future clinical trial to treat people hospitalized with influenza.

DETAILED DESCRIPTION:
There is a concern that the influenza virus will become resistant to the standard of care, oseltamivir (commonly known as Tamiflu), as resistance to this medication has been observed in people infected with the seasonal influenza virus. Because of the possibility of drug resistance, additional treatment options for influenza are needed. The purpose of this study is to collect blood from people who have recovered from influenza or who have received a seasonal influenza vaccine. The blood will then be processed into Food and Drug Administration (FDA)-licensed fresh frozen plasma (FFP). In a future clinical trial, this plasma will be used as a treatment for people hospitalized with influenza.

This study will enroll people who have recovered from influenza or received a seasonal influenza vaccine. Participants will donate blood at FDA-licensed blood donor centers up to three times during the 240-day study period.

ELIGIBILITY:
Inclusion Criteria:

* Currently healthy males 18 - 59 years of age with a history suggestive of having anti-influenza antibodies (either or both of the following):

  1. An influenza-like illness (e.g., fever, chills, malaise, cough, myalgias, nausea). Subjects must asymptomatic and must be afebrile for ≥ 7 days, and must enroll within 12 months of onset of illness.
  2. Vaccinated with a licensed influenza vaccine. Enrollment must occur >14 days and < 12 months from date of vaccination.
* Must be an adult male Department of Defense (DoD)/beneficiary
* Sign informed consent and Health Insurance Portability and Accountability Act (HIPAA) document
* A demonstrated H1N1 HAI titer of 1:160 or greater and H3N2 HAI titer of 1:40 or greater.
* Must also meet all Standard-of-Care inclusion criteria for donation of blood or plasma at the FDA-licensed donor center prior to every donation session. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Donors that do not meet all Standard-of-Care FDA approved requirements for the donation of blood and production of FFP as determined by the FDA-licensed donor center prior to every donation session may be excluded from further participation in this study. Study exclusion will be determined by the principal investigator (PI) or lead investigator at the study site.
* Donors that fail the Standard-of-Care screening and Blood Borne Pathogen screening for the following blood borne pathogens at the donor center will be excluded:

  1. Anti-HIV-I/II
  2. Anti-human T-lymphotropic virus (HTLV)-I/II
  3. Anti-hepatitis C (HCV)
  4. Anti-hepatitis B core antigen (HBc)
  5. Anti-T. cruzi (enzyme immunoassay [EIA] for Chagas disease) (if required by the FDA-licensed donor center or becomes a nationwide FDA requirement)
  6. Hepatitis B surface antigen (HBsAg)
  7. Serologic test for syphilis
  8. HIV nucleic acid test (NAT)
  9. HCV NAT
  10. West Nile virus (WNV) NAT
* Participation in other medical research that includes:

  1. Studies that are currently ongoing or will start during the duration of this study that require more than 60 mL of blood to be donated in any 56-day period of time
  2. Administration of any unlicensed drug in the 3 months before study entry or during the duration of this study
  3. Administration of any unlicensed vaccine in the 12 months before study entry or during the duration of this study, with the exception of unlicensed influenza vaccine

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will include people who have recovered from influenza, received a seasonal influenza vaccine, or have both recovered from influenza and received a seasonal influenza vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-04; Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Collection of high antibody titer anti-influenza FFP | Collected at each study visit

SECONDARY OUTCOMES:
Further define the hemagglutination inhibition (HAI) immune response in participants over time | Collected at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: LCDR Nicholas Martin, USN, MSC, Principal Investigator — Virology and Rickettsial Diseases Department, Naval Medical Research Center
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Naval Medical Research Center, Bethesda, Maryland

REFERENCES:
- [Background] Kash JC, Qi L, Dugan VG, Jagger BW, Hrabal RJ, Memoli MJ, Morens DM, Taubenberger JK. Prior infection with classical swine H1N1 influenza viruses is associated with protective immunity to the 2009 pandemic H1N1 virus. Influenza Other Respir Viruses. 2010 May 1;4(3):121-7. doi: 10.1111/j.1750-2659.2010.00132.x. PMID 20409208
- [Background] Tang JW, Shetty N, Lam TT. Features of the new pandemic influenza A/H1N1/2009 virus: virology, epidemiology, clinical and public health aspects. Curr Opin Pulm Med. 2010 May;16(3):235-41. doi: 10.1097/MCP.0b013e3283375727. PMID 20375785